CLINICAL TRIAL: NCT01079676
Title: A Phase III, Non-inferiority Study Comparing Two Filgrastim Preparations in Preventing Chemotherapy Induced Neutropenia in Breast Cancer
Brief Title: A Non-inferiority Study Comparing Two Filgrastim Preparations in Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EF-026
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-10

CONDITIONS: Neutropenia in Breast Cancer
MeSH Terms: interventions — Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Filgrastim (Experimental)
  Interventions: Drug: Filgrastim (Eurofarma)
- Granulokine (Active Comparator)
  Interventions: Drug: Filgrastim (Granulokine, Amgen)

INTERVENTIONS:
Drug: Filgrastim (Eurofarma) — Filgrastim will be given at the daily dose of 5 µg/kg body weight, subcutaneously. The weight considered will be the actual weight, for patients weighing up to 120 kg.
  Arms: Filgrastim
Drug: Filgrastim (Granulokine, Amgen) — Granulokine will be given at the daily dose of 5 µg/kg body weight, subcutaneously. The weight considered will be the actual weight, for patients weighing up to 120 kg.
  Arms: Granulokine

SUMMARY:
This study primary objective and endpoints are compare the efficacy of two products containing filgrastim, evaluating if the formulation produced by Eurofarma can be considered non-inferior to the reference product.

DETAILED DESCRIPTION:
This study primary objective and endpoints are compare the efficacy of two products containing filgrastim, evaluating if the formulation produced by Eurofarma can be considered non-inferior to the reference product. For this, the study primary endpoint will be the rate of grade 4 neutropenia after the first cycle of chemotherapy, according to the classification Common Terminology Criteria for Adverse Events (CTC-AE).

The study secondary objectives will be to compare other efficacy aspects, as well as the tolerability of the two products containing filgrastim.

The secondary endpoints considered for the study will be:

* The febrile neutropenia rate;
* The rate of any grade 4 neutropenia;
* The duration of the grade 4 neutropenia;
* The frequency of the adverse events and the laboratory changes.

ELIGIBILITY:
Inclusion Criteria:

* Signed ICF;
* Diagnosis confirmed by anatomic pathology examination (cytology or histopathology) of breast cancer;
* Clinical or imaging confirmation of stage II to IV disease, according to the TNM classification;
* Indication for chemotherapy with one of the eligible regimens, as long as the treatment in the first cycle is planned as full dose (without adjustments relative to the original regimen);
* Performance status from 0 to 1 on the Zubrod scale;
* No more than one previous chemotherapeutic regimen for metastatic disease;
* Proper organic functions, as indicated by all the following conditions:

  * ANC >1500/mm3;
  * Platelet count >150000/mm3;
  * Serum creatinine <1,2 mg/dL;
  * Bilirubins and transaminases (aspartate aminotransferase [AST] and alanine aminotransferase [ALT]) <1.5 times the upper limit of normal.

Exclusion Criteria:

* Forecast of prophylactic or therapeutic use of antibiotics, antifungal or antiviral in the first cycle of chemotherapy;
* Previous radiotherapy involving pelvis or radiotherapy of any site on the last 6 weeks before randomization;
* History of bone marrow transplantation (as receptor);
* Presence of other neoplasias, with the exception of in situ cervical carcinoma, in situ bladder carcinoma, cutaneous basal cell carcinoma properly treated, cutaneous spinocellular carcinoma properly treated, T1 vocal cords cancer under remission or previous malignant neoplasia treated more than 5 years before the recruitment and without relapse;
* Presence of severe comorbidities, such as cardiovascular, chronic respiratory, kidney, liver, neurological, hematological, infectious, skin, neurological or psychiatric disease;
* Recent (< 12 months) or foreseen participation during this study in other clinical studies involving any nature of drugs or studies of any kind of intervention, unless there may be a direct benefit to the research subject, as per CNS/MS Resolution 251/97, item III.j.
* Intolerability or allergy to any of the components of the filgrastim formulations evaluated in the study.
* Pregnancy or lactation (patients of childbearing potential must have a negative blood pregnancy test on the 7 days prior to the randomization).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2011-03; Primary Completion 2011-04 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
The study primary endpoint will be the rate of grade 4 neutropenia after the first cycle of chemotherapy, according to the classification Common Terminology Criteria for Adverse Events (CTC-AE) | 5 months

SECONDARY OUTCOMES:
The febrile neutropenia rate. | 5 months

CONTACTS AND LOCATIONS:
Locations (6):
- Brazil (6):
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceição, Porto Alegre, Rio Grande do Sul
  - CEPHO - Faculdade de Medicina do ABC, Santo André, São Paulo
  - Casa de Saúde Santa Marcelina, São Paulo, São Paulo
  - Centro de Referência da Saúde da Mulher, São Paulo, São Paulo
  - IAVC - Instituto de Cancer Arnaldo Vieira de Carvalho, São Paulo, São Paulo